CLINICAL TRIAL: NCT01078220
Title: A Post-licensure Surveillance Program for the Safety of GARDASIL™ in a Managed Care Organization Setting
Brief Title: Observational Surveillance Study to Detect Potential Safety Signals in Patients Who Have Had at Least One Dose of GARDASIL™ (V501-031)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: V501-031; 2010_019; EP08014.031 (Other: Merck)
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Human Papillomavirus Infection
Keywords: Human Papillomavirus (HPV)
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 3-Dose Safety Population (Primary): Females between ages 9 to 26 at receipt of the first dose of GARDASIL who are members of the participating MCOs and have completed the 3-dose regimen of GARDSIL vaccination with 12 months.
- Pregnancy Safety Population: Females who received at least one dose of GARDASIL during pregnancy.
- Autoimmune Safety Population: Females who have received at least one dose of GARDASIL and have been members in the same MCO for at least 12 months prior to receiving their first dose of GARDASIL.
- Any Dose Safety Population (Secondary): Females who have received at least one dose of GARDASIL and have been members in the same MCO for at least 12 months prior to receiving their first dose of GARDASIL.

SUMMARY:
This is a post-licensure safety surveillance program to detect potential safety signals in subjects, from the managed care organizations database, who have used GARDASIL™.

ELIGIBILITY:
Inclusion Criteria:

3-Dose Safety Population

* Female 9-26 years at the time of first dose of GARDASIL™
* Completed the 3-dose regimen of GARDASIL™ per protocol

Pregnancy Safety Population

* Received at least one dose of GARDASIL™ up to 30 days prior to the date of conception or any time between conception and the day of pregnancy resolution

Autoimmune Safety Population

* Female who has received at least one dose of GARDASIL™
* Has been a member of same Managed Care Organization (MCO) for at least 12 months prior to the receipt of GARDASIL™

Any Dose Safety Population

* Female who has received at least one dose of GARDASIL™

Exclusion Criteria:

3-Dose Safety Population

* Male
* Receives incomplete regimen of GARDASIL™
* Completes the three dose regimen of GARDASIL™ in more than 12 months
* Less than 28 day interval between doses 1 and 2 or less than a 12 week interval between doses 2 and 3
* Younger than 9 or older than 26 years of age at receipt of first dose

Pregnancy Safety Population

* Males
* No record of pregnancy at the Managed Care Organization (MCO)

Autoimmune Safety Population

* Member of the same MCO for less than 12 months prior to receiving the first dose
* Male

Min Age: 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Managed Care Organizations (MCO) databases
Sampling Method: Probability Sample
Enrollment: 189629 (Actual)
Dates: Start 2007-02-06 (Actual); Primary Completion 2010-12-13 (Actual); Study Completion 2010-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Chao C, Klein NP, Velicer CM, Sy LS, Slezak JM, Takhar H, Ackerson B, Cheetham TC, Hansen J, Deosaransingh K, Emery M, Liaw KL, Jacobsen SJ. Surveillance of autoimmune conditions following routine use of quadrivalent human papillomavirus vaccine. J Intern Med. 2012 Feb;271(2):193-203. doi: 10.1111/j.1365-2796.2011.02467.x. Epub 2011 Nov 15. PMID 21973261
- [Result] Klein NP, Hansen J, Chao C, Velicer C, Emery M, Slezak J, Lewis N, Deosaransingh K, Sy L, Ackerson B, Cheetham TC, Liaw KL, Takhar H, Jacobsen SJ. Safety of quadrivalent human papillomavirus vaccine administered routinely to females. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1140-8. doi: 10.1001/archpediatrics.2012.1451. PMID 23027469
- See also: EUPAS Register (EUPAS17730) — http://www.encepp.eu/encepp/viewResource.htm?id=17731

RESULTS

PARTICIPANT FLOW:
Groups:
- Any Dose Safety Population: Any female who received any dose of Gardasil at a managed care organization (MCO) between August 2006 and March 2008.
Period: Overall Study
Arm/Group | Any Dose Safety Population
Started | 189629
Completed | 189629
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Any Dose Safety Population
Number analyzed (Participants) | 189629
Age, Customized [Number; unit: Participants]
  <9 years | 45
  Between 9 and 15 years | 96839
  Between 16 and 26 years | 91066
  >26 years | 1679
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189629
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Syncope
Description: Syncope was defined as the presence of a syncope diagnosis code in the emergency room or hospital setting in the vaccination risk period or in the post-vaccination self-comparison period. These codes could have represented a new event, a pre-existing event, a prior history of the event, a "rule out" diagnosis, miscoding, or a misdiagnosis. Consistent with the study's design, diagnosis codes for general safety analyses were not confirmed in this study.
Time Frame: On day of each vaccination
Measure: Number; unit: Rate per 1000 person years
Groups:
- Any Dose Safety Population: Any female who received any dose of Gardasil at a MCO between August 2006 and March 2008.
- 3-Dose Safety Population: Any female who was 9-26 years old at first dose of Gardasil and who was a MCO member at each dose, and who had a minimum of 28 days between doses 1 and 2, and 12 weeks between doses 2 and 3, and who received all 3 doses of Gardasil within 12 months
Arm/Group | Any Dose Safety Population | 3-Dose Safety Population
Number analyzed (Participants) | 189629 | 44001
Rate per 1000 person years | 24.21 | 13.84
Statistical Analysis 1: Comparison: Any Dose Safety Population; Test type: Superiority or Other; unconditional logistic regression; Relative Risk = 6.00, 95% CI 2-sided [3.91 to 9.21] — Relative risk was approximated by odds ratio, obtained from conditional logistic regression
Statistical Analysis 2: Comparison: 3-Dose Safety Population; Test type: Superiority or Other; unconditional logistic regression; Relative Risk = 2.88, 95% CI 2-sided [1.18 to 7.08] — Relative risk was approximated by odds ratio, obtained from conditional logistic regression

2. Secondary Outcome: Number of Congenital Anomalies Among Females Who Received Gardasil During Pregnancy
Description: Pregnancy exposure was defined as receipt of Gardasil at any time from 1 month prior to conception through end of pregnancy.
Time Frame: First dose of Gardasil in pregnancy up to 6 months after birth
Population: Number of females potentially exposed to Gardasil during potential pregnancy as identified from unconfirmed diagnosis codes in electronic medical records.
Measure: Number; unit: Number of congenital anomalies
Groups:
- Pregnancy Safety Population: Any female from the Any Dose Safety Population with suspected exposure to Gardasil during pregnancy.
Arm/Group | Pregnancy Safety Population
Number analyzed (Participants) | 1740
Number of congenital anomalies
  Number (No.) of potential congenital anomalies | 170
  No. that underwent medical record review | 170
  No. of confirmed congenital anomalies | 44
  No. associated with Gardasil by safety committee | 0

3. Secondary Outcome: Number of Miscarriages Among Females Who Received Gardasil During Pregnancy
Description: as for outcome 2
Time Frame: First dose of Gardasil in pregnancy up to pregnancy resolution
Population: as for outcome 2
Measure: Number; unit: Number of miscarriages
Arm/Group | Pregnancy Safety Population
Number analyzed (Participants) | 1740
Number of miscarriages
  No. of potential miscarriages indentified | 633
  No. that underwent medical record review | 100
  No. of confirmed miscarriages | 9
  No. associated with Gardasil by safety committee | 0

4. Secondary Outcome: Number of Cases of New Onset Autoimmune Conditions in Females Receiving at Least One Dose of Gardasil
Description: Autoimmune cases were defined as newly diagnosed cases within 6 months after any
  dose of Gardasil, as confirmed by medical record review by panels of physicians specializing in the 16 autoimmune conditions of interest.
Time Frame: within 6 months immediately after each vaccination
Population: Number of females with at least 12 months' membership at a MCO prior to Gardasil.
Measure: Number; unit: Number of autoimmune cases
Groups:
- Autoimmune Safety Population: Any female with at least 12 months of membership at a MCO prior to their first dose of Gardasil, in order to exclude pre-existing conditions prior to their first dose of Gardasil.
Arm/Group | Autoimmune Safety Population
Number analyzed (Participants) | 149306
Number of autoimmune cases
  No. of potential autoimmune cases | 719
  No. that underwent medical record review | 318
  No. of confirmed new onset cases within 6 months | 124
  No. associated with Gardasil by safety committee | 0

5. Primary Outcome: Incidence Rate of Cellulitis
Description: Cellulitis was defined as the presence of a cellulitis or abscess diagnosis code in the emergency room or hospital setting in the vaccination risk period or in the post-vaccination self-comparison period. These codes could have represented a new event, a pre-existing event, a prior history of the event, a "rule out" diagnosis, miscoding, or a misdiagnosis. Consistent with the study's design, diagnosis codes for general safety analyses were not confirmed in this study.
Time Frame: Within 14 days and within 60 days immediately after each vaccination
Measure: Number; unit: Rate per 1000 person years
Arm/Group | Any Dose Safety Population | 3-Dose Safety Population
Number analyzed (Participants) | 189629 | 44001
Rate per 1000 person years
  Days 1-14 after vaccination | 3.53 | 2.17
  Days 1-60 after vaccination | 2.25 | 1.66
Statistical Analysis 1: Comparison: Any Dose Safety Population; Days 1-14 after vaccination; Test type: Superiority or Other; unconditional logistic regression; Relative Risk = 1.64, 95% CI 2-sided [1.17 to 2.3] — Relative risk was approximated by odds ratio, obtained from conditional logistic regression
Statistical Analysis 2: Comparison: Any Dose Safety Population; Days 1-60 after vaccination; Test type: Superiority or Other; unconditional logistic regression; Relative Risk = 1.05, 95% CI 2-sided [0.82 to 1.35] — Relative risk was approximated by odds ratio, obtained from conditional logistic regression
Statistical Analysis 3: Comparison: 3-Dose Safety Population; Days 1-14 after vaccination; Test type: Superiority or Other; unconditional logistic regression; Relative Risk = 1.02, 95% CI 2-sided [0.53 to 1.98] — Relative risk was approximated by odds ratio, obtained from conditional logistic regression
Statistical Analysis 4: Comparison: 3-Dose Safety Population; Days 1-60 after vaccination; Test type: Superiority or Other; unconditional logistic regression; Relative Risk = 0.78, 95% CI 2-sided [0.5 to 1.21] — Relative risk was approximated by odds ratio, obtained from conditional logistic regression

ADVERSE EVENTS:
Description: Per protocol, non-serious adverse events and serious adverse events (SAEs)
  were not required to be captured as part of the study database, therefore, none were collected, and the number at risk is zero.
Arm/Group | Any Dose Safety Population
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Details of syncope and cellulitis findings and null findings for hundreds of other general safety analyses will be described in future publications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.